CLINICAL TRIAL: NCT03944369
Title: A Randomized, Open-Label, Prospective, Parallel Group, 2-Part Clinical Food Study to Assess the Safety, Tolerability, and Effect of KB109 on the Gut Microbiome in Subjects Whose Gastrointesinal Tracts Are Colonized With Multiple Drug-resistant Organisms
Brief Title: VITORA: Clinical Study to Evaluate the Effect of KB109 on the Gut Microbiome in Subjects Whose Gastrointestinal Tracts Are Colonized With Multiple Drug-resistant Organisms
Acronym: VITORA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K017-119
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Vancomycin-Resistant Enterococcus, Extended-Spectrum Beta Lactamase-Producing Enterobacteriaceae, or Carbapenem-Resistant Enterobacteriaceae Colonized Subjects
Keywords: Microbiome; Antibiotic resistance; Carbapenem-Resistant Enterobacteriaceae (CRE); Extended-Spectrum Beta Lactamase-Producing Enterobacteriaceae (ESBLE); Vancomycin-resistant Enterococcus (VRE); Multi Drug Resistant Organism (MDRO); Drug resistant; Kaleido; VITORA; KB109; Microbiome Metabolic Therapy (MMT); Oligosaccharide; Glycan

STUDY DESIGN:
Intervention Model Description: A Randomized, Open-Label, Prospective, Parallel Group, 2-Part Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational Control (Other): The observational control arm is an observational control group.
  Interventions: Other: No intervention
- KB109 (Other): KB109 is a novel glycan.
  Interventions: Other: KB109

INTERVENTIONS:
Other: KB109 — KB109 is a novel glycan
  Arms: KB109
Other: No intervention — No intervention
  Arms: Observational Control

SUMMARY:
This randomized, open-label, clinical study aims to explore the safety and tolerability of KB109, a novel glycan, versus an observational control group on the gut microbiome in subjects whose gastrointestinal tracts are colonized with multiple drug-resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, ≥18 years of age
* Positive stool culture for at least one of these three organisms: VRE, ESBLE or CRE
* Be willing and able to give informed consent
* If taking probiotic or prebiotic dietary supplements, usage must be consistent within 7 days prior to the run-in phase and willing to remain consistent throughout the study
* If subject is female: subject is surgically sterile or post-menopausal (12 months with no menses without an alternate medical cause); or if subject is a female of childbearing potential, must have a negative urine pregnancy test at Screening, must not be lactating, and must agree to abstain from sexual activity or agree to use one highly effective method of contraception for the duration of the study

Exclusion Criteria:

* Planned escalation of immunosuppression
* Neutropenia (≤500 absolute neutrophil count per μL)
* Allogenic stem cell transplant recipients with ongoing gastrointestinal disease
* Rapidly progressive or terminal illness
* Hemodynamic instability, or any other significant systemic, unstable or untreated disease
* Currently receiving or anticipated to require systemic (oral or IV anti-infective) or gut-directed antibacterial therapy
* Recent history of the following conditions requiring medical attention: known or suspected gastrointestinal (GI) infection (e.g., viral or bacterial gastroenteritis) or inflammatory bowel disease
* Major intra-abdominal surgery related to the bowel within the 3 months prior to Run-In
* Receiving total parenteral nutrition
* Contraindications, sensitivity, or known allergy to the use of the study product or its components
* Individuals who, in the opinion of the Investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study procedures (e.g., planned procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of product-related treatment-emergent adverse events (TEAEs) | Day -7 through Day 42
Incidence of serious adverse events (SAEs) | Day -7 through Day 42
Change in Bristol Stool Scale (BSS) through the collection of daily patient questionnaires. | Day -7 through Day 42]
  Evaluate the effect of KB109 on self-report questionnaires including the Bristol Stool Scale, an assessment of stool consistency on a scale from 1 (separate hard lumps, like nuts, hard to pass) through 7 (watery, no solid pieces, entirely liquid)

SECONDARY OUTCOMES:
1. Proportion of subjects with a reduction from baseline on Day 28 in the relative abundance of taxa of interest (Enterobacteriaceae, Enterococcus, and C. difficile, individually) as measured by metagenomic sequencing. | Day -1 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Boisciences
Locations (8):
- United States (8):
  - Harbor UCLA Medical Center, Torrance, California
  - Emory University, Atlanta, Georgia
  - Augusta Universtiy, Augusta, Georgia
  - Newland Immunology Center of Excellence; Providence Hospital, Southfield, Michigan
  - Stony Brook University, Stony Brook, New York
  - Atrium Health's Carolinas Medical Center, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas